CLINICAL TRIAL: NCT05449509
Title: Association of SYNTAX Score With Abdominal Aortic Aneurysm in Patients Undergoing Coronary Artery Bypass Graft Surgery: Who Should be Screened?
Brief Title: Abdominal Aortic Aneurysm Screening Before Coronary Artery Bypass Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Kamile Özeren Topçu, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Other Study IDs: KAEK/2022.02.43
Record Dates: First submitted 2022-07-02; First posted 2022-07-08 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Coronary Artery Disease; Abdominal Aortic Aneurysm
MeSH Terms: conditions — Coronary Artery Disease; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-SYNTAX score patients
  Interventions: Diagnostic Test: Abdominal aortic Duplex ultrasound
- Intermediate/low-SYNTAX score patients
  Interventions: Diagnostic Test: Abdominal aortic Duplex ultrasound

INTERVENTIONS:
Diagnostic Test: Abdominal aortic Duplex ultrasound — All patients will undergo bedside Duplex ultrasound in order to measure infrarenal abdominal aortic diameter.

SUMMARY:
Coronary artery disease (CAD) and abdominal aortic aneurysm (AAA) are two separate entities with common risk factors such as hypertension, advanced age, male sex. Atherosclerosis plays an important role in the etiology of both diseases. It has been reported that AAA is more prevalent in patients undergoing coronary artery bypass grafting (CABG). Despite all the evidence, current guidelines do not recommend routine screening for AAA before CABG. Syntax score shows anatomical significance of CAD and is associated with the degree of atherosclerotic load. The investigators aim to investigate if there were any differences regarding AAA prevalence in high-SYNTAX patients versus intermediate/low-SYNTAX patients.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing coronary artery bypass graft surgery
* Age >18 years

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Breastfeeding
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients undergoing elective CABG in the Department of Cardiovascular Surgery in Basaksehir Cam Sakura City Hospital
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Infrarenal abdominal aortic diameter | Baseline
  Infrarenal abdominal aortic diameter measured by bedside Duplex ultrasound by the principal investigator, Dr. Ozeren-Topcu

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam ve Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergersen L, Kiernan MS, McFarlane G, Case TD, Ricci MA. Prevalence of abdominal aortic aneurysms in patients undergoing coronary artery bypass. Ann Vasc Surg. 1998 Mar;12(2):101-5. doi: 10.1007/s100169900124. PMID 9514225
- [Background] Yammine M, Itagaki S, Pawale A, Toyoda N, Reddy RC. SYNTAX score may predict the severity of atherosclerosis of the ascending aorta. J Thorac Dis. 2017 Oct;9(10):3859-3865. doi: 10.21037/jtd.2017.09.17. PMID 29268395